CLINICAL TRIAL: NCT04839367
Title: Positron Emission Tomography Imaging of Participants With Confirmed Prostate Cancer Using 64Cu-SAR-bisPSMA: A Multi-Centre, Blinded Review, Dose Ranging Phase I Study
Brief Title: Positron Emission Tomography (PET) Imaging of Participants With Confirmed Prostate Cancer Using 64Cu-SAR-bisPSMA (PROPELLER)
Acronym: PROPELLER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP03
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 - 100 MBq 64Cu-SAR-bisPSMA (Experimental): Participants will receive a single administration, a bolus injection of 100 MBq 64Cu-SAR-bisPSMA.
  Interventions: Drug: 64Cu-SAR-bisPSMA
- Cohort 2 - 150 MBq 64Cu-SAR-bisPSMA (Experimental): Participants will receive a single administration, a bolus injection of 150 MBq 64Cu-SAR-bisPSMA.
  Interventions: Drug: 64Cu-SAR-bisPSMA
- Cohort 3 - 200 MBq 64Cu-SAR-bisPSMA (Experimental): Participants will receive a single administration, a bolus injection of 200 MBq 64Cu-SAR-bisPSMA.
  Interventions: Drug: 64Cu-SAR-bisPSMA

INTERVENTIONS:
Drug: 64Cu-SAR-bisPSMA — 64Cu-SAR-bisPSMA

SUMMARY:
The aim of this study is to determine the safety and tolerability of 64Cu-SARbisPSMA in participants with untreated, confirmed Prostate Cancer.

DETAILED DESCRIPTION:
This is a multi-centre, blinded review, dose ranging, non-randomized study of 64Cu-SAR-bisPSMA administered to participants with confirmed Prostate Cancer. 30 eligible participants will be allocated (1:1:3) to 1 of 3 dosing cohorts to be administered with 64Cu-SAR-bisPSMA 100 MBq, 150 MBq or 200 MBq. PET/CT scan images will be sent to blinded central readers to assess the capacity of 64Cu-SAR-bisPSMA to detect primary Prostate Cancer, to assess image quality of the various dose cohorts, and to assess the PET/CT scan features of 64Cu-SAR-bisPSMA in comparison standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* ≥18 years of age;
* Life expectancy >3 months;
* Confirmation of Prostate Cancer by histopathology and planned radical prostatectomy;
* Have ≥1 of the following intermediate- to high-risk features:

  1. PSA level greater than or equal to 10.0 ng/ml within 12 weeks prior to enrolment;
  2. International Society of Urological Pathology (ISUP) Grade Group 3 (i.e. Gleason score of 7 (4+3) or above;
  3. Clinical stage greater than or equal to T2b;
* Participants must have adequate renal function;
* Sexually active participants who have female partners of childbearing potential: Partner and/or participant must agree to use an acceptable form of contraception. Further participants must refrain from donating sperm;
* A 68Ga-PSMA-11 PET/CT scan performed within 5 weeks, but not closer than 6 hours prior to the administration of 64Cu-SAR-bisPSMA.

Exclusion Criteria:

* Prior prostatectomy or any other treatment for Prostate Cancer, including Androgen Deprivation Therapy and radiation therapy;
* Previous treatment with PSMA-targeted therapy within 3 months prior to enrolment, and administration of other investigational agents within 4 weeks prior to entering the study (except 68Ga-PSMA-11);
* Known hypersensitivity to the components of 64Cu-SAR-bisPSMA;
* Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, participants with a prior history of malignancy that has been adequately treated and who have been disease free for more than 3 years are eligible, as are participants with adequately treated non-melanoma skin cancer, superficial bladder cancer;
* Any serious medical condition which the Investigator feels may interfere with the procedures or evaluations of the study;
* Patients unwilling or unable to comply with protocol or with a history of noncompliance or inability to grant informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 64Cu-SAR-bisPSMA using Common Terminology Criteria for Adverse Events version 5 | 11 weeks
  Safety will be assessed via vital signs, pathology tests (hematology, biochemistry, urinalysis, coagulation), physical examinations, ECGs and spontaneous AE reporting.
Efficacy of 64Cu-SAR-bisPSMA in the Detection of Primary Prostate Caner Compared to Histopathology | 11 weeks
  Efficacy will be measured by the proportion of 64Cu-SAR-bisPSMA PET/CT scans assessed as True Positive or False Negative for primary Prostate Cancer, as confirmed by histopathology.

SECONDARY OUTCOMES:
Comparison of image quality at varying dose levels of 64CuSAR-bisPSMA for each dose cohort (100 MBq, 150 MBq and 200 MBq). | 11 weeks
  Image quality will be assessed by 2 blinded central readers.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - GenesisCare CTA, SJOG Medical Clinic, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No